CLINICAL TRIAL: NCT00947518
Title: Does Skin Cleansing With Chlorhexidine Affect Skin Condition, Temperature and Colonization in Hospitalized Preterm Low Birth Weight Infants?: A Randomized Clinical Trial
Brief Title: Safety of Skin Cleansing With Chlorhexidine in Preterm Low Birth Weight Infants
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: All India Institute of Medical Sciences (Other)
Responsible Party: M Jeeva Sankar, Department of Pediatrics, AIIMS, New Delhi
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 10/2004
Record Dates: First submitted 2009-04-20; First posted 2009-07-28 (Estimated); Results first posted 2009-07-28 (Estimated); Last update posted 2018-06-25 (Actual); Status verified 2009-06

CONDITIONS: Neonatal Sepsis; Low Birth Weight
Keywords: chlorhexidine; preterm; newborn; skin condition; temperature; skin flora
MeSH Terms: conditions — Neonatal Sepsis; Premature Birth; Skin Diseases | interventions — Chlorhexidine; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Chlorhexidine skin cleansing (Experimental): Wiping the skin (except the face) once immediately after birth using baby wipes containing 0.25% free chlorhexidine (equivalent to 0.44% chlorhexidine digluconate)
  Interventions: Drug: Chlorhexidine
- Saline skin cleansing (Placebo Comparator): Wiping the skin (except the face) once immediately after birth using baby wipes containing normal saline
  Interventions: Drug: Normal saline
- No skin cleansing (No Intervention): No skin application

INTERVENTIONS:
Drug: Chlorhexidine — Baby wipes containing 0.25% free chlorhexidine (equivalent to 0.44% chlorhexidine digluconate)
  Arms: Chlorhexidine skin cleansing
Drug: Normal saline — Cleansing the skin (except the face)with baby wipes containing normal saline
  Arms: Saline skin cleansing

SUMMARY:
The purpose of this study is to examine if single skin cleansing with 0.25% chlorhexidine affects skin condition, temperature, and bacterial colonization in stable preterm (28-36 weeks gestational age) low birth weight (1001-2000 g) infants admitted in a health facility.

DETAILED DESCRIPTION:
Infections are the leading cause of death in neonates admitted to hospital - studies from developing countries suggest that about 25-71% of deaths occurring in neonatal intensive care units are secondary to infections.Such high infection-related mortality mandates an urgent implementation of simple and effective measures to prevent the occurrence of infections in these units.

The majority of neonatal infections occur in the first two weeks of life, when the epidermal barrier is immature and functionally compromised. Topical application of antiseptics until the skin matures could theoretically prevent skin colonization and reduce the incidence of systemic infections in neonates. Chlorhexidine, a broad-spectrum antiseptic used frequently for umbilical cord care in neonates, is now being evaluated for topical application to the skin. Hospital-based studies, involving predominantly term infants, have shown reductions in skin flora8 and a reduction in the incidence of sepsis following topical chlorhexidine application. In a community-based study in Nepal, a single skin cleansing with 0.25% chlorhexidine resulted in reduction in mortality among low birth weight infants; though the mechanism of the impact could not be determined, it was presumably due to increased susceptibility to transcutaneous sepsis in the low birth weight group.

Since the risk of infection in neonates is inversely related to their gestation, it is essential to evaluate the effect and the mechanism of such intervention in preterm neonates. These infants are, however, more prone to develop skin reactions following use of topical antiseptics. Preterm infants are also more prone to develop hypothermia following bathing/cleansing with antiseptic solution(s).

Since few studies have evaluated the effects of topical application of chlorhexidine in preterm infants admitted in a health care facility, we conducted the present study to examine if single skin cleansing with 0.25% chlorhexidine immediately after birth affects skin condition, temperature, and colonization in hospitalized preterm low birth weight infants.

ELIGIBILITY:
Inclusion Criteria:

* Preterm infants of 28 to 36 weeks' gestation
* Birth weights between 1001 and 2000 g

Exclusion Criteria:

* Infants with one minute Apgar score < 4
* Hemodynamic instability
* Congenital malformations
* Generalized skin disorder and
* Infants who need respiratory support (continuous positive airway pressure and/or intermittent mandatory ventilation) in the first 2-3 hours of life

Ages: 1 Hour to 3 Hours | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 60 (Actual)
Dates: Start 2005-08; Primary Completion 2006-02 (Actual); Study Completion 2006-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mari J Sankar, MD DM, Principal Investigator — Department of Pediatrics, All India Institute of Medical Sciences, New Delhi; Vinod K Paul, MD PhD, Study Chair — Department of Pediatrics, All India Institute of Medical Sciences, New Delhi; Ashok K Deorari, MD MNAMS, Study Chair — Department of Pediatrics, All India Institute of Medical Sciences, New Delhi; Gary L Darmstadt, MD MS, Study Chair — Department of International Health, Bloomberg School of Public Health, Johns Hopkins University

RESULTS

PARTICIPANT FLOW:
Recruitment Details: from August 2005 to February 2006 at the tertiary level neonatal intensive care unit of All India Institute of Medical Sciences, New Delhi
Pre-assignment Details: Infants with one minute Apgar score <4, hemodynamic instability, congenital malformations, generalized skin disorder and who needed respiratory support (continuous positive airway pressure and/or intermittent mandatory ventilation) were excluded
Groups:
- Chlorhexidine Skin Cleansing: Wiping the skin (except the face) using baby wipes containing 0.25% free chlorhexidine (equivalent to 0.44% chlorhexidine digluconate)
- Saline Skin Cleansing: Wiping the skin (except the face) using baby wipes containing normal saline
Period: Overall Study
Arm/Group | Chlorhexidine Skin Cleansing | Saline Skin Cleansing | No Skin Cleansing
Started | 20 | 20 | 20
Completed | 20 | 20 | 20
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Chlorhexidine Skin Cleansing | Saline Skin Cleansing | No Skin Cleansing | Total
Number analyzed (Participants) | 20 | 20 | 20 | 60
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 20 | 20 | 20 | 60
  Between 18 and 65 years | 0 | 0 | 0 | 0
  >=65 years | 0 | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 11 | 11 | 29
  Male | 13 | 9 | 9 | 31
Gestation (weeks) [Median (Full Range); unit: weeks] — Estimated gestational age in completed weeks
  weeks | 33 [28 to 36] | 33 [28 to 36] | 32.5 [28 to 36] | 33 [28 to 36]

OUTCOME MEASURES:

1. Primary Outcome: Median Skin Condition Score on the 9-point Skin Condition Grading Scale Adapted by Darmstadt From Lane et al
Description: The skin condition grading scale assesses the condition of the skin on the abdomen and dorsum of the hands/feet based on drying, erythema, crusting, oozing, etc. on a continuous scale from 1 (normal) to 9 (vesicles or pustules)
Time Frame: At 24 hours
Measure: Median (Full Range); unit: score on a scale
Arm/Group | Chlorhexidine Skin Cleansing | Saline Skin Cleansing | No Skin Cleansing
Number analyzed (Participants) | 20 | 20 | 20
score on a scale | 1 [1 to 2] | 1 [1 to 3] | 1 [1 to 2]
Statistical Analysis 1: Comparison: Chlorhexidine Skin Cleansing vs Saline Skin Cleansing vs No Skin Cleansing; Test type: Superiority or Other; p = 0.99, Kruskal-Wallis

2. Primary Outcome: Skin Temperature at 30 Min After Intervention
Description: Axillary skin temperature measured by a clinical thermometer kept in axilla for 3 minutes
Time Frame: at 30 min after intervention
Measure: Mean (Standard Deviation); unit: Degree Celsius
Arm/Group | Chlorhexidine Skin Cleansing | Saline Skin Cleansing | No Skin Cleansing
Number analyzed (Participants) | 20 | 20 | 20
Degree Celsius | 36.6 (0.2) | 36.6 (0.12) | 36.7 (0.24)
Statistical Analysis 1: Comparison: Chlorhexidine Skin Cleansing vs Saline Skin Cleansing vs No Skin Cleansing; Test type: Superiority or Other; p = 0.46, ANOVA

3. Primary Outcome: Number of Participants With Positive Skin Culture at Axilla
Description: Occurrence of any bacterial flora irrespective of the colony count in the skin swabs from axilla at 24 hrs after intervention
Time Frame: 24 hours after intervention
Measure: Number; unit: participants
Arm/Group | Chlorhexidine Skin Cleansing | Saline Skin Cleansing | No Skin Cleansing
Number analyzed (Participants) | 18 | 19 | 19
participants | 4 | 10 | 11
Statistical Analysis 1: Comparison: Chlorhexidine Skin Cleansing vs Saline Skin Cleansing vs No Skin Cleansing; Test type: Superiority or Other; p = 0.06, Chi-squared

4. Secondary Outcome: Incidence of Clinical and Culture Positive Sepsis
Description: Infants with symptoms and/or signs suggestive of sepsis and a positive blood culture (with known pathogens and coagulase negative staphylococcus) were diagnosed to have culture positive sepsis; Those with negative cultures but with positive sepsis screen were classified as having clinical sepsis
Time Frame: First week of life
Measure: Count of Participants; unit: Participants
Arm/Group | Chlorhexidine Skin Cleansing | Saline Skin Cleansing | No Skin Cleansing
Number analyzed (Participants) | 20 | 20 | 20
Participants
  Culture-positive sepsis | 1 | 2 | 2
  Clinical sepsis | 2 | 3 | 1
Statistical Analysis 1: Comparison: Chlorhexidine Skin Cleansing vs Saline Skin Cleansing vs No Skin Cleansing; Test type: Superiority; p < 0.05, Chi-squared; For comparison of categorical variables among the three groups, Chi2 test followed by Bonferroni's correction was used

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No